CLINICAL TRIAL: NCT04493931
Title: A Pharmacokinetic, Multi-cohort Study in Healthy Adult Subjects to Assess Gepotidacin as Victim and as Perpetrator of Drug-Drug Interactions Via CYP450, Renal and Intestinal Transporters, and to Assess Gepotidacin Pharmacokinetics in Japanese Healthy Adults
Brief Title: Drug-drug Interaction Study of Gepotidacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 213678
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Infections, Bacterial
Keywords: Gepotidacin; Drug Interaction; Pharmacokinetic; Safety; Bacterial Infection; Japanese Healthy Adults
MeSH Terms: conditions — Bacterial Infections | interventions — gepotidacin; Cimetidine; Rifampin; Midazolam; Digoxin

STUDY DESIGN:
Intervention Model Description: Cohort 1 and 2 are open-label, fixed sequence DDI cohorts. Cohort 3 is an open-label, 2-sequence, 2-period crossover randomized DDI cohort. Cohort 4 is a double-blind, placebo-controlled, randomized sequence study to investigate the safety and PK of gepotidacin.
Who Masked: Participant, Investigator
Masking Description: Cohort 1 to 3 are open-label cohorts. Cohort 4 is a double-blind cohort which contains blinded treatment of gepotidacin and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg (Experimental): This is a fixed sequence (Sequence AB) cohort. Participants will receive gepotidacin 1500 milligrams (mg) single dose (SD) on Day 1 of Period 1 (Treatment A); and Cimetidine 400 mg 4 times daily on Days 1 through 4 of Period 2 and gepotidacin 1500 mg single dose (Treatment B). Gepotidacin will be administered 1 hour after the first dose of cimetidine on Day 2 of Period 2. There will be a washout of at least 3 days between Treatment A and Treatment B, and a follow-up visit 5 to 7 days after the last dose of cimetidine.
  Interventions: Drug: Gepotidacin; Drug: Cimetidine
- Cohort 2: Gepotidacin 1500 mg + Rifampicin 600 mg (Experimental): This is a fixed sequence (Sequence CDE) cohort. Participants will receive gepotidacin 1500 mg single dose on Day 1 of Period 1 (Treatment C), rifampicin 600 mg (administered in the evenings) once daily for 7 days (Days 1 through 7 of Period 2, to elicit maximal enzyme induction) (Treatment D); and gepotidacin 1500 mg single dose administered in the morning on Day 8 and rifampicin 600 mg administered in the evening on Days 8 and 9 of Period 2 (Treatment E). There will be a washout of at least 3 days between Treatment C and Treatment D, and a follow-up visit 7 to 10 days after the last dose of rifampicin.
  Interventions: Drug: Gepotidacin; Drug: Rifampicin
- Cohort 3: Digoxin 0.5mg+Midazolam 2mg then Gepotidacin 3000mg (Experimental): Participants will receive digoxin 0.5 mg and midazolam 2 mg (Treatment F) in Period 1 on Day 1 then gepotidacin two 3000 mg doses (given 12 hours apart) co-administered with digoxin 0.5 mg and midazolam 2 mg in Period 2 on Day 1, with the 2 probe drugs administered with the second daily dose of gepotidacin only (Treatment G). There will be a washout of at least 10 days between treatments. In Sequence 2, these regimens are reversed. A follow-up visit will occur 7 to 10 days after the last dose of study intervention in Period 2.
  Interventions: Drug: Gepotidacin; Drug: Midazolam; Drug: Digoxin
- Cohort 3: Gepotidacin 3000mg then Digoxin 0.5mg+Midazolam 2mg (Experimental): Participants will receive gepotidacin two 3000 mg doses (given 12 hours apart) co-administered with digoxin 0.5 mg and midazolam 2 mg in Period 1 on Day 1, with the 2 probe drugs administered with the second daily dose of gepotidacin only (Treatment G) followed by digoxin 0.5 mg and midazolam 2 mg (Treatment F) in Period 2 on Day 1. A follow-up visit will occur 7 to 10 days after the last dose of study intervention in Period 2.
  Interventions: Drug: Gepotidacin; Drug: Midazolam; Drug: Digoxin
- Cohort 4: Gepotidacin 1500 mg fed then fasted then 3000 mg fed (Experimental): Cohort 4 will include Japanese participants. Participants will receive a single dose of gepotidacin 1500 mg under fed conditions in Period 1 (Treatment H), then a single dose of gepotidacin 1500 mg under fasted conditions in Period 2 (Treatment I), followed by two doses of gepotidacin up to 3000 mg (given 12 hours apart) under fed conditions in Period 3 (Treatment J). There will be a washout of at least 3 days between each treatment, and a follow-up visit 5 to 7 days after the last dose of gepotidacin.
  Interventions: Drug: Gepotidacin
- Cohort 4: Gepotidacin 1500 mg fasted then fed then 3000 mg fed (Experimental): Cohort 4 will include Japanese participants. Participants will receive a single dose of gepotidacin 1500 mg under fasted conditions in Period 1 (Treatment I), then a single dose of gepotidacin 1500 mg under fed conditions in Period 2 (Treatment H), followed by two doses of gepotidacin up to 3000 mg (given 12 hours apart) under fed conditions in Period 3 (Treatment J). There will be a washout of at least 3 days between each treatment, and a follow-up visit 5 to 7 days after the last dose of gepotidacin.
  Interventions: Drug: Gepotidacin
- Cohort 4: Placebo fed then fasted then fed (Placebo Comparator): Cohort 4 will include Japanese participants. Participants will receive a single dose of placebo under fed conditions in Period 1, then a single dose of placebo under fasted conditions in Period 2, followed by two doses of placebo (given 12 hours apart) under fed conditions in Period 3. There will be a washout of at least 3 days between each period, and a follow-up visit 5 to 7 days after the last dose of placebo.
  Interventions: Other: Placebo matching to gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin tablets will be available as unit dose strength 750 mg and will be administered orally.
  Other Names: GSK2140944
  Arms: Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Cohort 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Cohort 3: Digoxin 0.5mg+Midazolam 2mg then Gepotidacin 3000mg; Cohort 3: Gepotidacin 3000mg then Digoxin 0.5mg+Midazolam 2mg; Cohort 4: Gepotidacin 1500 mg fasted then fed then 3000 mg fed; Cohort 4: Gepotidacin 1500 mg fed then fasted then 3000 mg fed
Drug: Cimetidine — Cimetidine tablets will be available as unit dose strength 400 mg and will be administered orally.
  Arms: Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Drug: Rifampicin — Rifampicin Capsules will be available as unit dose strength 300 mg and will be administered orally.
  Arms: Cohort 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Drug: Midazolam — Midazolam oral syrup 2 milligrams per milliliter (mg/mL) will be available to be administered orally.
  Arms: Cohort 3: Digoxin 0.5mg+Midazolam 2mg then Gepotidacin 3000mg; Cohort 3: Gepotidacin 3000mg then Digoxin 0.5mg+Midazolam 2mg
Drug: Digoxin — Digoxin tablets will be available as unit dose strength 0.25 mg and will be administered orally.
  Arms: Cohort 3: Digoxin 0.5mg+Midazolam 2mg then Gepotidacin 3000mg; Cohort 3: Gepotidacin 3000mg then Digoxin 0.5mg+Midazolam 2mg
Other: Placebo matching to gepotidacin — Placebo matching to gepotidacin tablets will be administered orally.
  Arms: Cohort 4: Placebo fed then fasted then fed

SUMMARY:
This study is a drug-drug interaction (DDI), pharmacokinetics (PK), safety and tolerability study in adult healthy participants, including Japanese cohort. This study is designed to assess co-administration of probe substrates with gepotidacin in study cohorts 1 to 3 and establishing PK and safety in Japanese participants in cohort 4. Food effect will also be evaluated in cohort 4.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to (>=) 18 to less than or equal to (=<) 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead ECG results. A participant with clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Additional inclusion criteria for Japanese participants (Cohort 4): The participant is a non-naturalized Japanese citizen and holds a Japanese passport (current or expired).

The participant has/had 2 Japanese parents and 4 Japanese grandparents who are/were all non-naturalized Japanese citizens, as confirmed by interview.

The participant has been living outside of Japan for up to 10 years as confirmed by interview.

* Participants have a body weight >=40 kilograms (kg) and body mass index within the range 18.5 to 32.0 kilograms per square meter (kg/m^2) (inclusive).
* Male and/or female: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and 1 of the following conditions applies: Is a woman of non-childbearing potential or Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of <1 percent (%), for at least 30 days prior to dosing until completion of the follow-up Visit. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention.

A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) before the first dose of study intervention and for women not on effective contraception at least 14 days prior to baseline visit.

The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

* Clinically significant abnormality in the past medical history or at the screening physical examination that in the investigator's opinion may place the participant at risk or interfere with the outcome variables of the study. This includes, but is not limited to, history or current cardiac, hepatic, renal, neurologic, gastro-intestinal (GI), respiratory, hematologic, or immunologic disease.
* Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention, or any other condition that may place the participant at risk, in the opinion of the investigator.
* Female participant has a positive pregnancy test result or is lactating at Screening or upon admission to the clinic.
* Positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Note: Testing will be performed according to site procedures.
* Within 2 months before Screening, either a confirmed history of Clostridium difficile (C. difficile) diarrhea infection or a past positive of C. difficile toxin test.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of drug and/or alcohol abuse within 6 months before Screening, as determined by the investigator, or has a positive drug screen at Screening or upon admission to the clinic.
* History of sensitivity/hypersensitivity to any of the study drugs, components thereof, or a history of drug or other allergy that, in the opinion of the Investigator or GlaxoSmithKline (GSK) Medical Monitor contraindicates their participation.
* Cohort 2 Only: Participant is a contact lens wearer who is unable or unwilling to wear glasses for the duration of the study and for 5 half-lives after the last dose of rifampicin.
* Use of any systemic antibiotic within 30 days of screening.
* Participants must abstain from taking prescription or non-prescription drugs (except for hormonal contraceptives and/or acetaminophen at doses of <=2 grams/day), vitamins, and dietary or herbal supplements, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to study intervention until completion of the follow-up Visit, unless, in the opinion of the investigator and Sponsor, the medication will not interfere with the study. Any exceptions will be discussed with the Sponsor or Medical Monitor on a case-by-case basis and the reasons will be documented.
* Previous exposure to gepotidacin.
* Participant has participated in a clinical trial and has received an investigational product (IP) prior to gepotidacin administration within 30 days, 5 half-lives, or twice the duration of the biological effect of IP (whichever is longer).
* Past participation in this clinical study.
* Baseline corrected QT interval using the Fridericia formula (QTcF) of >450 milliseconds (msec) at Screening or Check-in.
* Presence of hepatitis B surface antigen or positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention.
* Alanine aminotransferase (ALT) >1.5 times upper limit of normal (ULN) at Screening or Check-in.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at Screening or Check-in.
* History of any kidney disease or current or chronic history of mild impaired renal function as indicated by an estimated creatinine clearance <=90 milliliters per minute (mL/min).
* A positive test for human immunodeficiency virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of Screening defined as an average weekly intake of >21 units (or an average daily intake of >3 units) for males or an average weekly intake of >14 units (or an average daily intake >2 units) for females. One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits, or 100 mL of wine.
* Cohort 3 Only: Digoxin-related exclusions include the following at Screening:

Serum potassium >5.5 milliequivalent per liter (mEq/L) or < 3.6 mEq/L Serum magnesium <1.6 milligrams per deciliter (mg/dL) Serum calcium (total) <8.5 mg/dL History of hypersensitivity to digoxin or other digitalis glycosides Any clinically relevant abnormality on 12-lead ECG at Screening or Check-in.

* Participant has donated blood in excess of 500 mL within 12 weeks prior to dosing or participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Participant is unable to comply with all study procedures, in the opinion of the investigator.
* Participant should not participate in the study, in the opinion of the investigator or Sponsor.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States and designed to assess co-administration of probe substrates with gepotidacin in study Cohorts 1 to 3 and establishing pharmacokinetics and safety in a Japanese cohort in Cohort 4.
Pre-assignment Details: A total of 64 participants (14 in Cohort 1, 17 in Cohort 2, 19 in Cohort 3 and 14 participants in Cohort 4) were enrolled in the study.
Groups:
- Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg: Participants received a single oral dose of gepotidacin 1500 milligrams (mg) on Day 1 of Period 1 followed by a washout of at least 3 days. In Period 2, participants were administered with cimetidine 400 mg 4 times daily on Days 1 through 4 of Period 2 along with a single dose of gepotidacin 1500 mg administered one hour after the first dose of cimetidine on Day 2 of Period 2. Participants had a follow-up of 7 days after the last dose of cimetidine.
- Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin: Participants received a single oral dose of gepotidacin 1500 mg on Day 1 of Period 1 followed by a washout of at least 3 days. In Period 2, participants received rifampicin 600 mg (administered in the evenings) once daily for 7 days (Days 1 through 7) along with a single dose of gepotidacin 1500 mg administered in the morning on Day 8 and rifampicin 600 mg administered in the evening on Days 8 and 9 of Period 2. Participants had a follow-up of 10 days after the last dose of rifampicin.
- Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam: Participants received digoxin 0.5 mg and midazolam 2 mg on Day 1 of Period 1 followed by a washout of 10 days. In Period 2, participants were administered with two doses of gepotidacin 3000 mg given 12 hours apart along with co-administration of digoxin 0.5 mg and midazolam 2 mg with the second dose of gepotidacin on Day 1 of Period 2. Participants had a follow-up of 10 days after the last dose of study treatment in Period 2.
- Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam: Participants received two doses of gepotidacin 3000 mg given 12 hours apart along with co-administration of digoxin 0.5 mg and midazolam 2 mg with the second dose of gepotidacin on Day 1 of Period 1 followed by a washout of 10 days. In Period 2, participants were administered with digoxin 0.5 mg and midazolam 2 mg on Day 1 of Period 2. Participants had a follow-up of 10 days after the last dose of study treatment in Period 2.
- Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed: Japanese participants received a single dose of gepotidacin 1500 mg under fed conditions on Day 1 of Period 1 followed by a washout of 3 days . In Period 2, participants were administered with a single dose of gepotidacin 1500 mg under fasted conditions on Day 1 of Period 2 followed by a washout of 3 days. In Period 3, participants were administered with two doses of gepotidacin 3000 mg (given 12 hours apart) under fed conditions on Day 1 of Period 3. Participants had a follow-up of 7 days after the last dose of gepotidacin.
- Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed: Japanese participants received a single dose of gepotidacin 1500 mg under fasted conditions on Day 1 of Period 1 followed by a a washout of 3 days. In Period 2, participants were administered with a single dose of gepotidacin 1500 mg under fed conditions on Day 1 of Period 2 followed by a washout of 3 days. In Period 3, participants were administered with two doses of gepotidacin 3000 mg (given 12 hours apart) under fed conditions on Day 1 of Period 3. Participants had a follow-up of 7 days after the last dose of gepotidacin.
- Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed: Japanese participants received a single dose of placebo matching gepotidacin under fed conditions on Day 1 of Period 1 followed by a a washout of 3 days. In Period 2, participants were administered with a single dose of placebo matching gepotidacin under fasted conditions on Day 1 of Period 2, followed by a washout of 3 days. In Period 3, participants were administered with two doses of placebo matching gepotidacin (given 12 hours apart) under fed conditions on Day 1 of Period 3. Participants had a follow-up of 7 days.
Period: Cohort1:Treatment Period 1(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 14 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 13 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1:Washout Period 1 (Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 13 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 13 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort1:Treatment Period 2(Up to 4 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 13 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 13 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1: Follow-up (Up to 7 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 13 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 13 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort2:Treatment Period 1(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 17 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 17 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2:Washout Period 1(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 17 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 17 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort2:Treatment Period2(Up to 10 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 17 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 14 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: Follow-up (Up to 10 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 14 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 14 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort3:Treatment Period 1(Up to 5 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 10 | 9 | 0 | 0 | 0
Completed | 0 | 0 | 9 | 9 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Cohort3:Washout Period 1(Up to 10 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 9 | 9 | 0 | 0 | 0
Completed | 0 | 0 | 9 | 9 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort3:Treatment Period 2(Up to 5 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 9 | 9 | 0 | 0 | 0
Completed | 0 | 0 | 9 | 9 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: Follow-up (Up to 10 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 9 | 9 | 0 | 0 | 0
Completed | 0 | 0 | 9 | 9 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort4:Treatment Period 1(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 0 | 0 | 6 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 6 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort4:Washout Period 1(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 0 | 0 | 6 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 6 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort4:Treatment Period 2(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 0 | 0 | 6 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 6 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort4:Washout Period 2(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 0 | 0 | 6 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 6 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort4:Treatment Period 3(Up to 3 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 0 | 0 | 6 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 6 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4: Follow-up (Up to 7 Days)
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed
Started | 0 | 0 | 0 | 0 | 6 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 6 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Gepotidacin 1500 mg/Cimetidine + Gepotidacin 1500 mg | Cohort 2: Gepotidacin 1500 mg/Gepotidacin 1500 mg + Rifampicin | Cohort 3: Digoxin+Midazolam/Gepotidacin 3000 mg + Digoxin + Midazolam | Cohort 3: Gepotidacin 3000 mg + Digoxin + Midazolam/Digoxin+Midazolam | Cohort 4:Gepotidacin 1500 mg Fed/Gepotidacin 1500 mg Fasted/Gepotidacin 3000 mg Fed | Cohort 4:Gepotidacin 1500 mg Fasted/Gepotidacin 1500 mg Fed/Gepotidacin 3000 mg Fed | Cohort 4: Placebo Fed/ Placebo Fasted/ Placebo Fed | Total
Number analyzed (Participants) | 14 | 17 | 10 | 9 | 6 | 5 | 3 | 64
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-64 years | 14 | 17 | 10 | 9 | 6 | 5 | 3 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 3 | 5 | 2 | 2 | 2 | 25
  Male | 7 | 13 | 7 | 4 | 4 | 3 | 1 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 8 | 7 | 6 | 5 | 0 | 0 | 0 | 26
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  WHITE | 4 | 5 | 4 | 4 | 0 | 0 | 0 | 17
  BLACK OR AFRICAN AMERICAN/WHITE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ASIAN(A)/BLACK OR AFRICAN AMERICAN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  JAPANESE HERITAGE(H)/EAST A H/SOUTH EAST A H | 0 | 2 | 0 | 0 | 6 | 5 | 3 | 16
  AMERICAN INDIAN OR ALASKA NATIVE/WHITE | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Maximum Observed Concentration (Cmax) of Gepotidacin in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric least square (LS) mean and 90 percent (%) confidence interval (CI) of the geometric LS means have been presented.
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hour, 2 Hours 30 minutes, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours, 36 Hours, 48 Hours Post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population comprised of all participants in the Pharmacokinetic Population (received at least 1 dose of study intervention and had at least 1 non-missing plasma or urine pharmacokinetic concentration) who received study intervention for whom valid and evaluable plasma or urine pharmacokinetic parameters were derived.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Micrograms per milliliter
Groups:
- Cohort 1: Gepotidacin 1500 mg: Participants received a single oral dose of gepotidacin 1500 mg on Day 1 of Period 1 in Cohort 1.
- Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg: Participants received cimetidine 400 mg 4 times daily on Days 1 through 4 of Period 2 along with a single dose of gepotidacin 1500 mg administered one hour after the first dose of cimetidine on Day 2 of Period 2 in Cohort 1.
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Micrograms per milliliter | 4.817 [4.006 to 5.793] | 4.548 [3.756 to 5.506]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of Geometric LS Mean = 0.944, 90% CI 2-sided [0.753 to 1.184]

2. Primary Outcome: Cohort 1: Time to Reach Maximum Observed Concentration (Tmax) of Gepotidacin in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours | 2.500 [1.00 to 4.00] | 2.500 [1.00 to 4.00]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Median Difference (Final Values) = -0.250, 90% CI 2-sided [-0.750 to 0.742] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

3. Primary Outcome: Cohort 1: Terminal Phase Half-life (t1/2) of Gepotidacin in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric LS mean and 90% CI of the geometric LS means have been presented.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours | 11.344 [10.282 to 12.516] | 12.415 [11.207 to 13.754]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of Geometric LS Mean = 1.094, 90% CI 2-sided [0.959 to 1.249]

4. Primary Outcome: Cohort 1: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to the Time of the Last Quantifiable Concentration (AUC [0-t]) of Gepotidacin in Plasma
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours*micrograms per milliliter | 20.3 [17.7 to 23.3] | 23.4 [20.4 to 26.9]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of Geometric LS Mean = 1.157, 90% CI 2-sided [1.059 to 1.265]

5. Primary Outcome: Cohort 1: AUC From Time 0 (Pre-dose) Extrapolated to Infinite Time (AUC[0-infinity]) of Gepotidacin in Plasma
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours* micrograms per milliliter
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours* micrograms per milliliter | 20.6 [18.0 to 23.6] | 23.9 [20.8 to 27.4]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of Geometric LS Mean = 1.158, 90% CI 2-sided [1.062 to 1.264]

6. Primary Outcome: Cohort 2: Cmax of Gepotidacin in Plasma
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Micrograms per milliliter
Groups:
- Cohort 2:Period 1: Gepotidacin 1500 mg: Participants received a single oral dose of gepotidacin 1500 mg on Day 1 of Period 1 in Cohort 2.
- Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg: Participants received rifampicin 600 mg (administered in the evenings) once daily for 7 days (Days 1 through 7) followed by a single dose of Gepotidacin 1500 mg administered in the morning on Day 8 and rifampicin 600 mg administered in the evening on Days 8 and 9 of Period 2 in Cohort 2.
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Micrograms per milliliter | 3.735 [3.209 to 4.347] | 2.728 [2.323 to 3.202]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Ratio of Geometric LS Mean = 0.730, 90% CI 2-sided [0.635 to 0.840]

7. Primary Outcome: Cohort 2: Lag Time Before Observation of Drug Concentrations (Tlag) of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours | 0.000 [0 to 1.00] | 0.000 [0 to 0.50]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.000] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

8. Primary Outcome: Cohort 2: Tmax of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours | 2.500 [1.00 to 6.00] | 2.000 [1.00 to 4.00]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Median Difference (Final Values) = -0.467, 90% CI 2-sided [-1.000 to 0.492] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

9. Primary Outcome: Cohort 2: AUC(0-t) of Gepotidacin in Plasma
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours*micrograms per milliliter | 19.0 [16.9 to 21.3] | 9.0 [8.0 to 10.2]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Ratio of Geometric LS Mean = 0.476, 90% CI 2-sided [0.433 to 0.525]

10. Primary Outcome: Cohort 2: AUC(0-infinity) of Gepotidacin in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric LS mean and 90 % CI of the geometric LS means have been presented.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours*micrograms per milliliter | 19.3 [17.2 to 21.7] | 9.3 [8.2 to 10.4]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Ratio of Geometric LS Mean = 0.478, 90% CI 2-sided [0.435 to 0.526]

11. Primary Outcome: Cohort 3: Cmax of Digoxin in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of digoxin was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric LS mean and 90 % CI of the geometric LS means have been presented.
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 24 Hours, 36 Hours, 48 Hours, 72 Hours, 96 Hours Post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Picograms per milliliter
Groups:
- Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg: Participants received digoxin 0.5 mg and midazolam 2 mg on Day 1 of Period 1 and Period 2 in Cohort 3.
- Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg: Participants received two doses of gepotidacin 3000 mg given 12 hours apart along with co-administration of digoxin 0.5 mg and midazolam 2 mg with the second dose of gepotidacin on Day 1 of Period 1 and Period 2 in Cohort 3.
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Picograms per milliliter | 1553.135 [1318.390 to 1829.676] | 2381.259 [2013.503 to 2816.185]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.533, 90% CI 2-sided [1.274 to 1.845]

12. Primary Outcome: Cohort 3: Tlag of Digoxin in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of digoxin was conducted using standard non-compartmental analysis.
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours | 0.000 [0 to 0] | 0.000 [0 to 0]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.000] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

13. Primary Outcome: Cohort 3: Tmax of Digoxin in Plasma
Description: as for outcome 12
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours | 2.000 [0.50 to 4.00] | 1.275 [0.50 to 4.00]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Median Difference (Final Values) = -0.500, 90% CI 2-sided [-1.000 to -0.233] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

14. Primary Outcome: Cohort 3: AUC(0-t) of Digoxin in Plasma
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*picograms per milliliter
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 17
Hours*picograms per milliliter | 25353.1 [22490.9 to 28579.6] | 30842.3 [27241.5 to 34919.0]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.217, 90% CI 2-sided [1.085 to 1.363]

15. Primary Outcome: Cohort 3: AUC(0-infinity) of Digoxin in Plasma
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*picograms per milliliter
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours*picograms per milliliter | 30743.6 [27425.5 to 34463.1] | 34456.5 [30652.1 to 38733.1]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.121, 90% CI 2-sided [0.983 to 1.278]

16. Primary Outcome: Cohort 3: Cmax of Midazolam in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of midazolam was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric LS mean and 90 % CI of the geometric LS means have been presented.
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours, 36 Hours, 48 Hours Post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Nanograms per milliliter | 5.238 [4.436 to 6.185] | 6.507 [5.492 to 7.711]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.242, 90% CI 2-sided [1.046 to 1.475]

17. Primary Outcome: Cohort 3: Tlag of Midazolam in Plasma
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of midazolam was conducted using standard non-compartmental analysis.
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours | 0.000 [0 to 0] | 0.000 [0 to 0]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.000] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

18. Primary Outcome: Cohort 3: Tmax of Midazolam in Plasma
Description: as for outcome 17
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours | 0.650 [0.50 to 2.50] | 0.500 [0.50 to 4.00]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [-0.250 to 0.800] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

19. Primary Outcome: Cohort 3: AUC(0-t) of Midazolam in Plasma
Description: as for outcome 16
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*nanograms per milliliter
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours*nanograms per milliliter | 23.3 [19.5 to 27.9] | 44.8 [37.4 to 53.8]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.923, 90% CI 2-sided [1.622 to 2.278]

20. Primary Outcome: Cohort 3: AUC(0-infinity) of Midazolam in Plasma
Description: as for outcome 16
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*nanograms per milliliter
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours*nanograms per milliliter | 24.9 [21.1 to 29.6] | 47.4 [39.9 to 56.4]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.902, 90% CI 2-sided [1.619 to 2.234]

21. Primary Outcome: Cohort 4: Cmax of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- Cohort 4: Gepotidacin 1500 mg Fed: Japanese participants received a single dose of gepotidacin 1500 mg under fed conditions on Day 1 of Period 1 and Period 2 in Cohort 4.
- Cohort 4: Gepotidacin 1500 mg Fasted: Japanese participants received a single dose of gepotidacin 1500 mg under fasted conditions on Day 1 of Period 1 and Period 2 in Cohort 4.
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Micrograms per milliliter | 5.436 (27.8) | 5.143 (34.2)

22. Primary Outcome: Cohort 4: Tmax of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours | 2.000 [1.50 to 4.00] | 1.500 [1.00 to 4.00]

23. Primary Outcome: Cohort 4: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to the Concentration at 24 Hours Post-dose (AUC[0-24]) of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hour, 2 Hours 30 minutes, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours*micrograms per milliliter | 20.9 (16.8) | 19.0 (12.9)

24. Primary Outcome: Cohort 4: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to the Concentration at 48 Hours Post-dose (AUC[0-48]) of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours*micrograms per milliliter | 21.9 (16.0) | 20.0 (13.2)

25. Primary Outcome: Cohort 4: AUC(0-t) of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours*micrograms per milliliter | 21.9 (16.0) | 20.0 (13.2)

26. Primary Outcome: Cohort 4: AUC(0-infinity) of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours*micrograms per milliliter | 22.3 (15.5) | 20.4 (13.3)

27. Primary Outcome: Cohort 4: Cmax of Gepotidacin in Plasma After the First Dose of 3000 mg -Fed State
Description: as for outcome 2
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3, 4, 6, 8, 12 Hours, 12 Hours 30 minutes, 13 Hours, 13 Hours 30 minutes, 14 Hours, 14 Hours 30 minutes, 15, 16, 18, 20, 24, 36, 48, 60 Hours post-dose in Treatment Period 3
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- Cohort 4: Gepotidacin 3000 mg Fed: Japanese participants received two doses of gepotidacin 3000 mg (given 12 hours apart) under fed conditions on Day 1 of Period 3 in Cohort 4.
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Micrograms per milliliter | 11.204 (45.0)

28. Primary Outcome: Cohort 4: Tmax of Gepotidacin in Plasma After the First Dose of 3000 mg -Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours | 2.000 [1.00 to 4.00]

29. Primary Outcome: Cohort 4: AUC From Time 0 (Predose) to Time Tau (AUC[0-tau]) of Gepotidacin in Plasma After the First Dose of 3000 Mg-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | 37.3 (25.4)

30. Primary Outcome: Cohort 4: Cmax of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Micrograms per milliliter | 12.363 (21.3)

31. Primary Outcome: Cohort 4: Tmax of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours | 2.000 [1.00 to 3.00]

32. Primary Outcome: Cohort 4: AUC(0-tau) of Gepotidacin in Plasma After the Second Dose of 3000 mg (Evening Dose)-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | 46.7 (23.1)

33. Primary Outcome: Cohort 4: Accumulation Ratio Based on Cmax (RoCmax) of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)-Fed State
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Accumulation ratio was calculated as Cmax after the second dose divided by Cmax after the first dose.
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Ratio | 1.103 (39.3)

34. Primary Outcome: Cohort 4: Accumulation Ratio Based on AUC(0-tau) (RoAUC) of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)-Fed State
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Accumulation ratio was calculated as AUC(0-tau) after the second dose, where 0 is the timepoint prior to second dose, divided by AUC(0-tau) after the first dose, where 0 is the predose timepoint prior to the first dose.
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Ratio | 1.254 (13.1)

35. Primary Outcome: Cohort 4: AUC(0-24) of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)-Fed State
Description: as for outcome 2
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3, 4, 6, 8, 12 Hours, 12 Hours 30 minutes, 13 Hours, 13 Hours 30 minutes, 14 Hours, 14 Hours 30 minutes, 15, 16, 18, 20, 24 Hours post-dose in Treatment Period 3
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | 84.6 (23.1)

36. Primary Outcome: Cohort 4: AUC(0-48) of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)-Fed State
Description: as for outcome 2
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3, 4, 6, 8, 12 Hours, 12 Hours 30 minutes, 13 Hours, 13 Hours 30 minutes, 14 Hours, 14 Hours 30 minutes, 15, 16, 18, 20, 24, 36, 48 Hours post-dose in Treatment Period 3
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | 90.8 (22.9)

37. Primary Outcome: Cohort 4: AUC(0-t) of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | 91.4 (23.0)

38. Primary Outcome: Cohort 4: Number of Participants With Serious Adverse Events (SAE) and Non-serious Adverse Events (Non-SAE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any serious adverse event that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situations as per Medical or scientific judgment.
Time Frame: Up to 22 days
Population: Safety Population comprised of all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 4: Placebo: Japanese participants received a single oral dose of placebo matching gepotidacin under fed conditions in Period 1 or a single dose of placebo matching gepotidacin under fasted conditions in Period 2 or two doses of placebo (given 12 hours apart) matching gepotidacin under fed conditions in Period 3 in Cohort 4.
- Cohort 4: Gepotidacin 3000 mg Fed: Japanese participants received two doses of gepotidacin 3000 mg (given 12 hours apart) under fed conditions on on Day 1 of Period 3 in Cohort 4.
Arm/Group | Cohort 4: Placebo | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 3 | 11 | 11 | 11
Participants
  Any SAE | 0 | 0 | 0 | 0
  Any non-SAE | 0 | 1 | 2 | 4

39. Primary Outcome: Cohort 4: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were collected at indicated time points for analysis of hematology parameters including Basophils, Eosinophils, Erythrocyte Mean Corpuscular Hemoglobin (MCH), Erythrocyte Mean Corpuscular Volume (MCV), Erythrocytes, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose laboratory (lab) value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 (%). High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 22 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 3 | 11 | 11 | 11
Participants
  Basophils; To Low | 0 | 0 | 0 | 0
  Basophils; To Normal or No Change | 3 | 11 | 9 | 10
  Basophils; To High | 0 | 0 | 2 | 1
  Eosinophils; To Low | 0 | 0 | 0 | 0
  Eosinophils; To Normal or No Change | 3 | 10 | 10 | 10
  Eosinophils; To High | 0 | 1 | 1 | 1
  MCH; To Low | 0 | 0 | 0 | 0
  MCH; To Normal or No Change | 3 | 11 | 11 | 11
  MCH; To High | 0 | 0 | 0 | 0
  MCV; To Low | 0 | 0 | 0 | 0
  MCV; To Normal or No Change | 2 | 10 | 10 | 9
  MCV; To High | 1 | 1 | 1 | 2
  Erythrocytes; To Low | 0 | 0 | 0 | 1
  Erythrocytes; To Normal or No Change | 3 | 10 | 11 | 10
  Erythrocytes; To High | 0 | 1 | 0 | 0
  Hematocrit; To Low | 0 | 0 | 0 | 0
  Hematocrit; To Normal or No Change | 3 | 10 | 11 | 10
  Hematocrit; To High | 0 | 1 | 0 | 1
  Hemoglobin; To Low | 0 | 0 | 0 | 0
  Hemoglobin; To Normal or No Change | 3 | 10 | 11 | 11
  Hemoglobin; To High | 0 | 1 | 0 | 0
  Leukocytes; To Low | 0 | 0 | 0 | 1
  Leukocytes; To Normal or No Change | 3 | 11 | 11 | 10
  Leukocytes; To High | 0 | 0 | 0 | 0
  Lymphocytes; To Low | 0 | 0 | 0 | 0
  Lymphocytes; To Normal or No Change | 3 | 11 | 11 | 11
  Lymphocytes; To High | 0 | 0 | 0 | 0
  Monocytes; To Low | 0 | 0 | 0 | 0
  Monocytes; To Normal or No Change | 3 | 11 | 11 | 11
  Monocytes; To High | 0 | 0 | 0 | 0
  Neutrophils; To Low | 0 | 0 | 1 | 1
  Neutrophils; To Normal or No Change | 3 | 11 | 10 | 10
  Neutrophils; To High | 0 | 0 | 0 | 0
  Platelets; To Low | 0 | 0 | 0 | 1
  Platelets; To Normal or No Change | 3 | 11 | 11 | 10
  Platelets; To High | 0 | 0 | 0 | 0

40. Primary Outcome: Cohort 4: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were collected at indicated time points for analysis of clinical chemistry parameters including Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase (Alk Phos), Aspartate Aminotransferase (AST), Bilirubin, Calcium, Carbon Dioxide, Chloride, Creatine Kinase, Creatinine, Direct Bilirubin, Glucose, Magnesium, Potassium, Protein, Sodium, Blood Urea Nitrogen (BUN). Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 22 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 3 | 11 | 11 | 11
Participants
  ALT; To Low | 0 | 0 | 0 | 0
  ALT; To Normal or No Change | 3 | 11 | 11 | 11
  ALT; To High | 0 | 0 | 0 | 0
  Albumin; To Low | 1 | 0 | 0 | 0
  Albumin; To Normal or No Change | 2 | 11 | 11 | 11
  Albumin; To High | 0 | 0 | 0 | 0
  Alk Phos; To Low | 0 | 0 | 0 | 0
  Alk Phos; To Normal or No Change | 3 | 11 | 11 | 11
  Alk Phos; To High | 0 | 0 | 0 | 0
  AST; To Low | 0 | 0 | 0 | 0
  AST; To Normal or No Change | 3 | 11 | 11 | 11
  AST; To High | 0 | 0 | 0 | 0
  Bilirubin; To Low | 0 | 0 | 0 | 0
  Bilirubin; To Normal or No Change | 2 | 11 | 11 | 11
  Bilirubin; To High | 1 | 0 | 0 | 0
  Calcium; To Low | 0 | 0 | 0 | 0
  Calcium; To Normal or No Change | 3 | 11 | 11 | 11
  Calcium; To High | 0 | 0 | 0 | 0
  Carbon Dioxide; To Low | 0 | 0 | 1 | 0
  Carbon Dioxide; To Normal or No Change | 3 | 11 | 10 | 11
  Carbon Dioxide; To High | 0 | 0 | 0 | 0
  Chloride; To Low | 0 | 0 | 0 | 0
  Chloride; To Normal or No Change | 3 | 11 | 11 | 11
  Chloride; To High | 0 | 0 | 0 | 0
  Creatine Kinase; To Low | 1 | 0 | 0 | 1
  Creatine Kinase; To Normal or No Change | 2 | 11 | 11 | 9
  Creatine Kinase; To High | 0 | 0 | 0 | 1
  Creatinine; To Low | 0 | 0 | 0 | 0
  Creatinine; To Normal or No Change | 3 | 11 | 11 | 11
  Creatinine;To High | 0 | 0 | 0 | 0
  Direct Bilirubin; To Low | 0 | 0 | 0 | 0
  Direct Bilirubin; To Normal or No Change | 2 | 11 | 11 | 11
  Direct Bilirubin; To High | 1 | 0 | 0 | 0
  Glucose; To Low | 0 | 0 | 0 | 0
  Glucose; To Normal or No Change | 3 | 11 | 11 | 11
  Glucose; To High | 0 | 0 | 0 | 0
  Magnesium; To Low | 0 | 0 | 0 | 0
  Magnesium; To Normal or No Change | 3 | 11 | 11 | 11
  Magnesium; To High | 0 | 0 | 0 | 0
  Potassium; To Low | 0 | 0 | 0 | 0
  Potassium; To Normal or No Change | 2 | 11 | 11 | 11
  Potassium; To High | 1 | 0 | 0 | 0
  Protein; To Low | 0 | 0 | 0 | 0
  Protein; To Normal or No Change | 3 | 11 | 11 | 11
  Protein; To High | 0 | 0 | 0 | 0
  Sodium; To Low | 0 | 0 | 0 | 0
  Sodium; To Normal or No Change | 3 | 11 | 11 | 11
  Sodium; To High | 0 | 0 | 0 | 0
  BUN; To Low | 0 | 0 | 0 | 0
  BUN; To Normal or No Change | 3 | 11 | 11 | 11
  BUN; To High | 0 | 0 | 0 | 0

41. Primary Outcome: Cohort 4: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Urine samples were collected at indicated time points for the analysis of urinalysis parameters including potential of hydrogen (pH) of urine, presence of glucose, protein, blood, ketones, bilirubin, nitrite, leukocyte esterase in urine by dipstick. Specific gravity of urine was measured by microscopic examination. Participants were counted in the worst case category that their value changes to (low, normal, high, or abnormal), unless there is no change in their category. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 22 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 3 | 11 | 11 | 11
Participants
  Bilirubin; To Normal or No Change | 3 | 11 | 11 | 11
  Bilirubin; To Abnormal | 0 | 0 | 0 | 0
  Glucose; To Normal or No Change | 3 | 11 | 11 | 11
  Glucose; To Abnormal | 0 | 0 | 0 | 0
  Ketones; To Normal or No Change | 2 | 11 | 11 | 11
  Ketones; To Abnormal | 1 | 0 | 0 | 0
  Leukocyte Esterase; To Normal or No Change | 2 | 9 | 11 | 9
  Leukocyte Esterase; To Abnormal | 1 | 2 | 0 | 2
  Nitrite; To Normal or No Change | 3 | 11 | 11 | 10
  Nitrite; To Abnormal | 0 | 0 | 0 | 1
  Occult Blood; To Normal or No Change | 2 | 11 | 10 | 10
  Occult Blood; To Abnormal | 1 | 0 | 1 | 1
  Protein; To Normal or No Change | 3 | 11 | 11 | 11
  Protein; To Abnormal | 0 | 0 | 0 | 0
  pH; To Low | 0 | 0 | 0 | 0
  pH; To Normal or No Change | 3 | 11 | 11 | 11
  pH; To High | 0 | 0 | 0 | 0
  Specific Gravity; To Low | 0 | 0 | 0 | 0
  Specific Gravity; To Normal or No Change | 3 | 11 | 11 | 11
  Specific Gravity; To High | 0 | 0 | 0 | 0

42. Primary Outcome: Cohort 4: Number of Participants With Worst Case Vital Sign Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate were measured in a semi-supine position after 5 minutes rest. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 22 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 3 | 11 | 11 | 11
Participants
  DBP; To Low | 0 | 1 | 0 | 0
  DBP; To Normal or No Change | 3 | 10 | 11 | 11
  DBP; To High | 0 | 0 | 0 | 0
  SBP; To Low | 0 | 1 | 1 | 0
  SBP; To Normal or No Change | 3 | 10 | 10 | 11
  SBP; To High | 0 | 0 | 0 | 0
  Pulse rate; To Low | 0 | 0 | 0 | 0
  Pulse rate; To Normal or No Change | 3 | 11 | 11 | 11
  Pulse rate; To High | 0 | 0 | 0 | 0

43. Primary Outcome: Cohort 4: Number of Participants With Any Increase in Maximum Post-Baseline Electrocardiogram (ECG) Parameter Corrected QT (QTc) Interval
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of at least 10 minutes using an ECG machine that automatically calculated the QTc interval. Number of participants with any increase of >450 milliseconds in corrected QT interval using the Bazett formula (QTcB) Interval and corrected QT interval using the Fridericia formula (QTcF) Interval has been reported.
Time Frame: Up to 22 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 3 | 11 | 11 | 11
Participants
  QTcB Interval | 1 | 8 | 3 | 9
  QTcF Interval | 1 | 1 | 0 | 2

44. Primary Outcome: Cohort 4: Cmax of Gepotidacin Following Single Dose of 1500 mg in Plasma - Food Effect in Japanese Participants
Description: as for outcome 10
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Micrograms per milliliter | 5.421 [4.610 to 6.374] | 5.158 [4.386 to 6.065]
Statistical Analysis 1: Comparison: Cohort 4: Gepotidacin 1500 mg Fed vs Cohort 4: Gepotidacin 1500 mg Fasted; Test type: Other; Ratio of geometric LS mean = 1.051, 90% CI 2-sided [0.824 to 1.340]

45. Primary Outcome: Cohort 4: Tlag of Gepotidacin Following Single Dose of 1500 mg in Plasma - Food Effect in Japanese Participants
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours | 0.000 [0 to 0.50] | 0.000 [0 to 0]
Statistical Analysis 1: Comparison: Cohort 4: Gepotidacin 1500 mg Fed vs Cohort 4: Gepotidacin 1500 mg Fasted; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.250] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

46. Primary Outcome: Cohort 4: Tmax of Gepotidacin Following Single Dose of 1500 mg in Plasma - Food Effect in Japanese Participants
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours | 2.000 [1.50 to 4.00] | 1.500 [1.00 to 4.00]
Statistical Analysis 1: Comparison: Cohort 4: Gepotidacin 1500 mg Fed vs Cohort 4: Gepotidacin 1500 mg Fasted; Test type: Other; Median Difference (Final Values) = 0.500, 90% CI 2-sided [-0.500 to 1.250] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

47. Primary Outcome: Cohort 4: AUC(0-t) of Gepotidacin Following Single Dose of 1500 mg in Plasma - Food Effect in Japanese Participants
Description: as for outcome 10
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*Micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours*Micrograms per milliliter | 21.9 [20.3 to 23.7] | 20.0 [18.5 to 21.6]
Statistical Analysis 1: Comparison: Cohort 4: Gepotidacin 1500 mg Fed vs Cohort 4: Gepotidacin 1500 mg Fasted; Test type: Other; Ratio of geometric LS mean = 1.094, 90% CI 2-sided [0.987 to 1.212]

48. Primary Outcome: Cohort 4: AUC(0-infinity) of Gepotidacin Following Single Dose of 1500 mg in Plasma - Food Effect in Japanese Participants
Description: as for outcome 10
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*Micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours*Micrograms per milliliter | 22.3 [20.7 to 24.1] | 20.4 [18.9 to 22.0]
Statistical Analysis 1: Comparison: Cohort 4: Gepotidacin 1500 mg Fed vs Cohort 4: Gepotidacin 1500 mg Fasted; Test type: Other; Ratio of geometric LS mean = 1.095, 90% CI 2-sided [0.991 to 1.209]

49. Secondary Outcome: Cohort 1: AUC (0-24) of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 23
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours*micrograms per milliliter | 19.3 (32.6) | 21.9 (29.7)

50. Secondary Outcome: Cohort 1: AUC(0-48) of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours*micrograms per milliliter | 20.3 (31.4) | 23.0 (28.4)

51. Secondary Outcome: Cohort 1: Tlag of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours | 0.000 [0 to 0.50] | 0.000 [0 to 0]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [-0.250 to 0.000] — The median difference and the 90% CI of the median difference were from Hodges-Lehmann estimate

52. Secondary Outcome: Cohort 1: Apparent Volume of Distribution (Vz/F) of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Liters | 1190.16 (34.0) | 1143.29 (30.6)

53. Secondary Outcome: Cohort 1: Apparent Oral Clearance (CL/F) of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Liters per Hour | 72.72 (31.2) | 64.14 (28.0)

54. Secondary Outcome: Cohort 1: Total Unchanged Drug (Ae Total) of Gepotidacin in Urine
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Ae total was calculated by adding all the fractions of drug collected over all the allotted time intervals. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric LS mean and 90 % CI of the geometric LS means have been presented.
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-24 Hours, 24-36 Hours, 36-48 Hours Post-dose in each Treatment periods 1 and 2
Population: as for outcome 14
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Milligrams
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 12 | 13
Milligrams | 337.92 [281.14 to 406.16] | 410.10 [343.16 to 490.08]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of geometric LS mean = 1.214, 90% CI 2-sided [1.000 to 1.473]

55. Secondary Outcome: Cohort 1: AUC(0-24) of Gepotidacin in Urine
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric LS mean and 90% CI of the geometric LS means have been presented.
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-24 Hours Post-dose in each Treatment periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours*micrograms per milliliter | 3292.1 [2639.2 to 4106.5] | 3612.4 [2888.5 to 4517.7]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of geometric LS mean = 1.097, 90% CI 2-sided [0.948 to 1.270]

56. Secondary Outcome: Cohort 1: AUC(0-48) of Gepotidacin in Urine
Description: as for outcome 55
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Hours*micrograms per milliliter | 3578.2 [2890.1 to 4430.0] | 3831.1 [3087.7 to 4753.4]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of geometric LS mean = 1.071, 90% CI 2-sided [0.939 to 1.221]

57. Secondary Outcome: Cohort 1: Renal Clearance (CLr) of Gepotidacin
Description: as for outcome 55
Time Frame: as for outcome 54
Population: as for outcome 14
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Liters per Hour
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 12 | 13
Liters per Hour | 16.06 [14.18 to 18.18] | 17.59 [15.62 to 19.81]
Statistical Analysis 1: Comparison: Cohort 1: Gepotidacin 1500 mg vs Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg; Test type: Other; Ratio of geometric LS mean = 1.096, 90% CI 2-sided [0.930 to 1.292]

58. Secondary Outcome: Cohort 1: Amount of Drug Excreted in Urine in a Time Interval (Ae[t1-t2]) of Gepotidacin
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Ae(t1-t2) measured the amount of drug excreted in urine at defined time intervals.
Time Frame: 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-24 Hours, 24-36 Hours, 36-48 Hours post-dose in each Treatment periods 1 and 2
Population: Pharmacokinetic Parameter Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Milligrams
  Ae (0-2), n=14, 13 | 28.66 (185.9) | NA (NA) — NA indicates that data was not available as urine concentrations were below the lower limit of quantification. Hence, data was not calculated.
  Ae (2-4), n=14, 12: number analyzed (Participants) | 14 | 12
  Ae (2-4), n=14, 12 | 89.18 (120.8) | 142.99 (42.7)
  Ae (4-6), n=14, 13 | 50.52 (119.1) | 82.77 (44.0)
  Ae (6-8); n=14, 13 | 34.38 (56.2) | 46.22 (55.3)
  Ae (8-12), n=12, 13: number analyzed (Participants) | 12 | 13
  Ae (8-12), n=12, 13 | 29.90 (38.3) | 30.97 (38.0)
  Ae (12-24), n=14, 13 | 25.44 (38.1) | 22.04 (121.3)
  Ae (24-36), n=14, 13 | 10.88 (43.1) | 8.76 (89.6)
  Ae (36-48), n=14, 13 | 4.50 (39.3) | 4.08 (88.5)

59. Secondary Outcome: Cohort 1: Percentage of the Given Dose of Drug Excreted in Urine (fe%) of Gepotidacin
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. fe% was calculated as: (Ae total divided by Dose) multiplied by 100 percent (%).
Time Frame: as for outcome 54
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 12 | 13
Percent dose excreted | 22.72 (53.2) | 26.90 (21.3)

60. Secondary Outcome: Cohort 1: Number of Participants With SAE and Non-SAE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any serious adverse event that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situations as per Medical or scientific judgment.
Time Frame: Up to 17 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Participants
  Any SAE | 0 | 0
  Any non-SAE | 0 | 0

61. Secondary Outcome: Cohort 1: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were collected at indicated time points for analysis of hematology parameters including Basophils, Eosinophils, MCH, MCV, Erythrocytes, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 %. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 17 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Participants
  Basophils; To Low | 0 | 0
  Basophils; To Normal or No Change | 14 | 11
  Basophils; To High | 0 | 2
  Eosinophils; To Low | 0 | 0
  Eosinophils; To Normal or No Change | 14 | 13
  Eosinophils; To High | 0 | 0
  MCH; To Low | 0 | 0
  MCH; To Normal or No Change | 14 | 13
  MCH; To High | 0 | 0
  MCV; To Low | 0 | 0
  MCV; To Normal or No Change | 13 | 13
  MCV; To High | 1 | 0
  Erythrocytes; To Low | 0 | 2
  Erythrocytes; To Normal or No Change | 14 | 11
  Erythrocytes; To High | 0 | 0
  Hematocrit; To Low | 0 | 1
  Hematocrit; To Normal or No Change | 13 | 12
  Hematocrit; To High | 1 | 0
  Hemoglobin; To Low | 0 | 0
  Hemoglobin; To Normal or No Change | 14 | 13
  Hemoglobin; To High | 0 | 0
  Leukocytes; To Low | 0 | 0
  Leukocytes; To Normal or No Change | 13 | 13
  Leukocytes; To High | 1 | 0
  Lymphocytes; To Low | 0 | 0
  Lymphocytes; To Normal or No Change | 14 | 12
  Lymphocytes; To High | 0 | 1
  Monocytes; To Low | 0 | 0
  Monocytes; To Normal or No Change | 13 | 13
  Monocytes; To High | 1 | 0
  Neutrophils; To Low | 0 | 1
  Neutrophils; To Normal or No Change | 13 | 12
  Neutrophils; To High | 1 | 0
  Platelets; To Low | 0 | 0
  Platelets; To Normal or No Change | 14 | 13
  Platelets; To High | 0 | 0

62. Secondary Outcome: Cohort 1: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were collected at indicated time points for analysis of clinical chemistry parameters including ALT, Albumin, Alk Phos, AST, Bilirubin, Calcium, Carbon Dioxide, Chloride, Creatine Kinase, Creatinine, Direct Bilirubin, Glucose, Magnesium, Potassium, Protein, Sodium, BUN. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 17 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Participants
  ALT; To Low | 0 | 0
  ALT; To Normal or No Change | 14 | 11
  ALT; To High | 0 | 2
  Albumin; To Low | 0 | 1
  Albumin; To Normal or No Change | 14 | 12
  Albumin; To High | 0 | 0
  Alk Phos; To Low | 0 | 0
  Alk Phos; To Normal or No Change | 14 | 13
  Alk Phos; To High | 0 | 0
  AST; To Low | 0 | 0
  AST; To Normal or No Change | 14 | 12
  AST; To High | 0 | 1
  Bilirubin; To Low | 0 | 1
  Bilirubin; To Normal or No Change | 14 | 12
  Bilirubin; To High | 0 | 0
  Calcium; To Low | 0 | 0
  Calcium; To Normal or No Change | 14 | 13
  Calcium; To High | 0 | 0
  Carbon Dioxide; To Low | 1 | 0
  Carbon Dioxide; To Normal or No Change | 13 | 13
  Carbon Dioxide; To High | 0 | 0
  Chloride; To Low | 0 | 0
  Chloride; To Normal or No Change | 14 | 12
  Chloride; To High | 0 | 1
  Creatine Kinase; To Low | 1 | 0
  Creatine Kinase; To Normal or No Change | 13 | 13
  Creatine Kinase; To High | 0 | 0
  Creatinine; To Low | 0 | 0
  Creatinine; To Normal or No Change | 14 | 10
  Creatinine; To High | 0 | 3
  Direct Bilirubin; To Low | 0 | 0
  Direct Bilirubin; To Normal or No Change | 14 | 13
  Direct Bilirubin; To High | 0 | 0
  Glucose; To Low | 0 | 0
  Glucose; To Normal or No Change | 14 | 13
  Glucose; To High | 0 | 0
  Magnesium; To Low | 0 | 0
  Magnesium; To Normal or No Change | 14 | 13
  Magnesium; To High | 0 | 0
  Potassium; To Low | 0 | 0
  Potassium; To Normal or No Change | 14 | 12
  Potassium; To High | 0 | 1
  Protein; To Low | 0 | 0
  Protein; To Normal or No Change | 14 | 13
  Protein; To High | 0 | 0
  Sodium; To Low | 0 | 0
  Sodium; To Normal or No Change | 14 | 13
  Sodium; To High | 0 | 0
  BUN; To Low | 0 | 0
  BUN; To Normal or No Change | 14 | 13
  BUN; To High | 0 | 0

63. Secondary Outcome: Cohort 1: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Urine samples were collected at indicated time points for the analysis of urinalysis parameters including pH of urine, presence of glucose, protein, blood, ketones, bilirubin, nitrite, leukocyte esterase in urine by dipstick. Specific gravity of urine was measured by microscopic examination. Participants were counted in the worst case category that their value changes to (low, normal, high, or abnormal), unless there is no change in their category. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 17 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Participants
  Bilirubin; To Normal or No Change | 14 | 13
  Bilirubin; To Abnormal | 0 | 0
  Glucose; To Normal or No Change | 14 | 13
  Glucose; To Abnormal | 0 | 0
  Ketones; To Normal or No Change | 14 | 13
  Ketones; To Abnormal | 0 | 0
  Leukocyte Esterase; To Normal or No Change | 12 | 13
  Leukocyte Esterase; To Abnormal | 2 | 0
  Nitrite; To Normal or No Change | 14 | 13
  Nitrite; To Abnormal | 0 | 0
  Occult Blood; To Normal or No Change | 13 | 11
  Occult Blood; To Abnormal | 1 | 2
  Protein; To Normal or No Change | 14 | 13
  Protein; To Abnormal | 0 | 0
  pH; To Low | 0 | 0
  pH; To Normal or No Change | 14 | 13
  pH; To High | 0 | 0
  Specific Gravity; To Low | 0 | 0
  Specific Gravity; To Normal or No Change | 13 | 13
  Specific Gravity; To High | 1 | 0

64. Secondary Outcome: Cohort 1: Number of Participants With Worst Case Vital Sign Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Vital signs including SBP, DBP and pulse rate were measured in a semi-supine position after 5 minutes rest. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 17 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Participants
  DBP; To Low | 0 | 0
  DBP; To Normal or No Change | 14 | 13
  DBP; To High | 0 | 0
  SBP; To Low | 0 | 0
  SBP; To Normal or No Change | 14 | 13
  SBP; To High | 0 | 0
  Pulse rate; To Low | 0 | 0
  Pulse rate; To Normal or No Change | 14 | 13
  Pulse rate; To High | 0 | 0

65. Secondary Outcome: Cohort 1: Number of Participants With Any Increase in Maximum Post-Baseline ECG Parameter QTc Interval
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of at least 10 minutes using an ECG machine that automatically calculated the QTc interval. Number of participants with any increase of >450 milliseconds in corrected QT interval using the QTcB Interval and QTcF Interval has been reported.
Time Frame: Up to 17 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg
Number analyzed (Participants) | 14 | 13
Participants
  QTcB Interval | 3 | 4
  QTcF Interval | 0 | 1

66. Secondary Outcome: Cohort 2: AUC(0-24) of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 23
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours*micrograms per milliliter | 17.9 (28.6) | 8.9 (29.6)

67. Secondary Outcome: Cohort 2: AUC(0-48) of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours*micrograms per milliliter | 19.0 (27.7) | 9.5 (28.5)

68. Secondary Outcome: Cohort 2: T1/2 of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours | 10.882 (25.5) | 10.972 (17.2)

69. Secondary Outcome: Cohort 2: Vz/F of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Liters | 1217.45 (37.0) | 2460.46 (39.2)

70. Secondary Outcome: Cohort 2: CL/F of Gepotidacin in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Liters per Hour | 77.55 (27.6) | 155.43 (27.9)

71. Secondary Outcome: Cohort 2: Ae Total of Gepotidacin in Urine
Description: as for outcome 54
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Milligrams
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Milligrams | 312.73 [286.95 to 340.82] | 156.05 [141.81 to 171.72]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Ratio of geometric LS mean = 0.499, 90% CI 2-sided [0.441 to 0.565]

72. Secondary Outcome: Cohort 2: AUC(0-24) of Gepotidacin in Urine
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed-effect model with treatment as a fixed effect and participant as a random effect. Geometric LS mean and 90 % CI of the geometric LS means have been presented.
Time Frame: as for outcome 55
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours*micrograms per milliliter | 3081.3 [2327.4 to 4079.5] | 1352.4 [1014.2 to 1803.4]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Ratio of geometric LS mean = 0.439, 90% CI 2-sided [0.370 to 0.521]

73. Secondary Outcome: Cohort 2: AUC(0-48) of Gepotidacin in Urine
Description: as for outcome 72
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Hours*micrograms per milliliter | 3370.1 [2571.4 to 4417.0] | 1476.8 [1119.2 to 1948.6]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Ratio of geometric LS mean = 0.438, 90% CI 2-sided [0.372 to 0.516]

74. Secondary Outcome: Cohort 2: CLr of Gepotidacin
Description: as for outcome 72
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Liters per Hour
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Liters per Hour | 16.49 [15.02 to 18.09] | 17.07 [15.47 to 18.84]
Statistical Analysis 1: Comparison: Cohort 2:Period 1: Gepotidacin 1500 mg vs Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg; Test type: Other; Ratio of geometric LS mean = 1.036, 90% CI 2-sided [0.950 to 1.129]

75. Secondary Outcome: Cohort 2: Ae(t1-t2) of Gepotidacin
Description: as for outcome 58
Time Frame: as for outcome 58
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Milligrams
  Ae (0-2) | 12.67 (567.5) | NA (NA) — NA indicates that data was not available as urine concentrations were below the lower limit of quantification. Hence, data was not calculated.
  Ae (2-4) | 79.84 (65.6) | 55.81 (47.4)
  Ae (4-6) | 67.48 (44.3) | 21.66 (66.4)
  Ae (6-8) | 33.92 (50.5) | 13.82 (56.1)
  Ae (8-12) | 27.59 (63.1) | 9.19 (50.7)
  Ae (12-24) | 21.17 (79.2) | 11.51 (36.4)
  Ae (24-36) | 11.04 (77.9) | 4.74 (42.7)
  Ae (36-48) | 3.61 (90.3) | 2.75 (31.8)

76. Secondary Outcome: Cohort 2: Percentage of the Given Dose of Drug Excreted in Urine (fe%) of Gepotidacin
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. fe% was calculated as: (Ae total divided by Dose) multiplied by 100 %.
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | Cohort 2:Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Percent dose excreted | 20.85 (16.9) | 10.42 (25.4)

77. Secondary Outcome: Cohort 2: Number of Participants With SAE and Non-SAE
Description: as for outcome 60
Time Frame: Up to 26 days
Population: Safety Population. Participants with adverse events that occurred during Days 1 to 7 in Period 2 after the exposure of rifampicin 600 mg and those occurred during Days 8 to 9 in Period 2 after exposure of gepotidacin 1500 mg + Rifampicin 600 mg were summarized separately. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Period 1: Gepotidacin 1500 mg: Participants received a single oral dose of gepotidacin 1500 mg on Day 1 of Period 1 in Cohort 2.
- Cohort 2: Period 2 (Days 1 to 7) Rifampicin 600 mg: Participants received rifampicin 600 mg (administered in the evenings) once daily for 7 days (Days 1 through 7) of Period 2 in Cohort 2.
- Cohort 2: Period 2 (Days 8 to 9) Gepotidacin 1500 mg + Rifampicin 600 mg: Participants received a single dose of gepotidacin 1500 mg administered in the morning on Day 8 and rifampicin 600 mg administered in the evening on Days 8 and 9 of Period 2 in Cohort 2.
Arm/Group | Cohort 2: Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2 (Days 1 to 7) Rifampicin 600 mg | Cohort 2: Period 2 (Days 8 to 9) Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 17 | 14
Participants
  Any SAE | 0 | 0 | 0
  Any non-SAE | 3 | 2 | 2

78. Secondary Outcome: Cohort 2: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were collected at indicated time points for analysis of hematology parameters including Basophils, Eosinophils, MCH, MCV, Erythrocytes, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 26 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 17
Participants
  Basophils; To Low | 0 | 0
  Basophils; To Normal or No Change | 17 | 16
  Basophils; To High | 0 | 1
  Eosinophils; To Low | 0 | 0
  Eosinophils; To Normal or No Change | 15 | 14
  Eosinophils; To High | 2 | 3
  MCH; To Low | 0 | 0
  MCH; To Normal or No Change | 17 | 17
  MCH; To High | 0 | 0
  MCV; To Low | 0 | 0
  MCV; To Normal or No Change | 17 | 17
  MCV; To High | 0 | 0
  Erythrocytes; To Low | 0 | 0
  Erythrocytes; To Normal or No Change | 17 | 17
  Erythrocytes; To High | 0 | 0
  Hematocrit; To Low | 0 | 0
  Hematocrit; To Normal or No Change | 14 | 15
  Hematocrit; To High | 3 | 2
  Hemoglobin; To Low | 0 | 0
  Hemoglobin; To Normal or No Change | 17 | 17
  Hemoglobin; To High | 0 | 0
  Leukocytes; To Low | 0 | 1
  Leukocytes; To Normal or No Change | 17 | 16
  Leukocytes; To High | 0 | 0
  Lymphocytes; To Low | 0 | 0
  Lymphocytes; To Normal or No Change | 17 | 15
  Lymphocytes; To High | 0 | 2
  Monocytes; To Low | 1 | 3
  Monocytes; To Normal or No Change | 15 | 14
  Monocytes; To High | 1 | 0
  Neutrophils; To Low | 0 | 4
  Neutrophils; To Normal or No Change | 17 | 13
  Neutrophils; To High | 0 | 0
  Platelets; To Low | 0 | 0
  Platelets; To Normal or No Change | 17 | 16
  Platelets; To High | 0 | 1

79. Secondary Outcome: Cohort 2: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 62
Time Frame: Up to 26 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 17
Participants
  ALT; To Low | 0 | 0
  ALT; To Normal or No Change | 17 | 15
  ALT; To High | 0 | 2
  Albumin; To Low | 0 | 0
  Albumin; To Normal or No Change | 17 | 17
  Albumin; To High | 0 | 0
  Alk Phos; To Low | 0 | 0
  Alk Phos; To Normal or No Change | 17 | 17
  Alk Phos; To High | 0 | 0
  AST; To Low | 0 | 0
  AST; To Normal or No Change | 17 | 16
  AST; To High | 0 | 1
  Bilirubin; To Low | 0 | 2
  Bilirubin; To Normal or No Change | 17 | 15
  Bilirubin; To High | 0 | 0
  Calcium; To Low | 0 | 0
  Calcium; To Normal or No Change | 17 | 17
  Calcium; To High | 0 | 0
  Carbon Dioxide; To Low | 0 | 3
  Carbon Dioxide; To Normal or No Change | 17 | 14
  Carbon Dioxide; To High | 0 | 0
  Chloride; To Low | 0 | 0
  Chloride; To Normal or No Change | 17 | 17
  Chloride; To High | 0 | 0
  Creatine Kinase; To Low | 0 | 0
  Creatine Kinase; To Normal or No Change | 17 | 17
  Creatine Kinase; To High | 0 | 0
  Creatinine; To Low | 0 | 0
  Creatinine; To Normal or No Change | 16 | 16
  Creatinine; To High | 1 | 1
  Direct Bilirubin; To Low | 0 | 0
  Direct Bilirubin; To Normal or No Change | 17 | 17
  Direct Bilirubin; To High | 0 | 0
  Glucose; To Low | 0 | 0
  Glucose; To Normal or No Change | 17 | 16
  Glucose; To High | 0 | 1
  Magnesium; To Low | 0 | 0
  Magnesium; To Normal or No Change | 17 | 17
  Magnesium; To High | 0 | 0
  Potassium; To Low | 0 | 0
  Potassium; To Normal or No Change | 16 | 15
  Potassium; To High | 1 | 2
  Protein; To Low | 0 | 0
  Protein; To Normal or No Change | 17 | 17
  Protein; To High | 0 | 0
  Sodium; To Low | 0 | 0
  Sodium; To Normal or No Change | 17 | 17
  Sodium; To High | 0 | 0
  BUN; To Low | 0 | 0
  BUN; To Normal or No Change | 17 | 17
  BUN; To High | 0 | 0

80. Secondary Outcome: Cohort 2: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 63
Time Frame: Up to 26 days
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 16
Participants
  Bilirubin; To Normal or No Change | 17 | 16
  Bilirubin; To Abnormal | 0 | 0
  Glucose; To Normal or No Change | 17 | 16
  Glucose; To Abnormal | 0 | 0
  Ketones; To Normal or No Change | 17 | 16
  Ketones; To Abnormal | 0 | 0
  Leukocyte Esterase; To Normal or No Change | 16 | 14
  Leukocyte Esterase; To Abnormal | 1 | 2
  Nitrite; To Normal or No Change | 17 | 15
  Nitrite; To Abnormal | 0 | 1
  Occult Blood; To Normal or No Change | 17 | 14
  Occult Blood; To Abnormal | 0 | 2
  Protein; To Normal or No Change | 17 | 16
  Protein; To Abnormal | 0 | 0
  pH; To Low | 0 | 0
  pH; To Normal or No Change | 17 | 16
  pH; To High | 0 | 0
  Specific Gravity; To Low | 0 | 0
  Specific Gravity; To Normal or No Change | 14 | 15
  Specific Gravity; To High | 3 | 1

81. Secondary Outcome: Cohort 2: Number of Participants With Worst Case Vital Sign Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 64
Time Frame: Up to 26 days
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Participants
  DBP; To Low | 0 | 0
  DBP; To Normal or No Change | 16 | 14
  DBP; To High | 1 | 0
  SBP; To Low | 0 | 0
  SBP; To Normal or No Change | 17 | 14
  SBP; To High | 0 | 0
  Pulse rate; To Low | 0 | 0
  Pulse rate; To Normal or No Change | 17 | 14
  Pulse rate; To High | 0 | 0

82. Secondary Outcome: Cohort 2: Number of Participants With Any Increase in Maximum Post-Baseline ECG Parameter QTc Interval
Description: as for outcome 65
Time Frame: Up to 26 days
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2: Gepotidacin 1500 mg + Rifampicin 600 mg
Number analyzed (Participants) | 17 | 14
Participants
  QTcB Interval | 2 | 2
  QTcF Interval | 0 | 1

83. Secondary Outcome: Cohort 3: Cmax of Gepotidacin in Plasma After the First Dose of 3000 mg (First Dose)
Description: as for outcome 2
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3, 4, 6, 8, 12 Hours, 12 Hours 30 minutes, 13 Hours, 13 Hours 30 Hours, 14 Hours, 14 Hours 30 Hours, 15, 16,18,20,24,36, 48, 60 Hours post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Micrograms per milliliter | 7.867 (36.8)

84. Secondary Outcome: Cohort 3: Tmax of Gepotidacin in Plasma After the First Dose of 3000 mg (First Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours | 2.500 [1.00 to 4.07]

85. Secondary Outcome: Cohort 3: Tlag of Gepotidacin in Plasma After the First Dose of 3000 mg (First Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours | 0.250 [0 to 1.00]

86. Secondary Outcome: Cohort 3: AUC(0-tau) of Gepotidacin in Plasma First Dose of 3000 mg (First Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours*micrograms per milliliter | 29.8 (30.8)

87. Secondary Outcome: Cohort 3: Cmax of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Micrograms per milliliter | 10.051 (47.7)

88. Secondary Outcome: Cohort 3: Tmax of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours | 2.000 [1.00 to 6.00]

89. Secondary Outcome: Cohort 3: AUC(0-tau) of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours* micrograms per milliliter | 41.9 (30.2)

90. Secondary Outcome: Cohort 3: RoCmax of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)
Description: as for outcome 33
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Ratio | 1.278 (54.4)

91. Secondary Outcome: Cohort 3: RoAUC of Gepotidacin in Plasma After the Second Dose of 3000 mg (Second Dose)
Description: as for outcome 34
Time Frame: as for outcome 83
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Ratio | 1.406 (27.5)

92. Secondary Outcome: Cohort 3: AUC(0-24) of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 2
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3, 4, 6, 8, 12 Hours, 12 Hours 30 minutes, 13 Hours, 13 Hours 30 Hours, 14 Hours, 14 Hours 30 Hours, 15, 16,18,20,24 Hours post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours*micrograms per milliliter | 73.2 (26.8)

93. Secondary Outcome: Cohort 3: AUC(0-48) of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 2
Time Frame: Pre-dose, 30 minutes, 1 Hour, 1 Hour 30 minutes, 2 Hours, 2 Hours 30 minutes, 3, 4, 6, 8, 12 Hours, 12 Hours 30 minutes, 13 Hours, 13 Hours 30 Hours, 14 Hours, 14 Hours 30 Hours, 15, 16,18,20,24,36, 48 Hours post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours*micrograms per milliliter | 81.2 (25.9)

94. Secondary Outcome: Cohort 3: AUC(0-t) of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 17
Hours*micrograms per milliliter | 85.2 (20.1)

95. Secondary Outcome: Cohort 3: Vz/F of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 17
Liters | 959.42 (30.0)

96. Secondary Outcome: Cohort 3: CL/F of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 17
Liters per Hour | 69.99 (20.1)

97. Secondary Outcome: Cohort 3: T1/2 of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose+ Second Dose)
Description: as for outcome 2
Time Frame: as for outcome 83
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 17
Hours | 9.501 (22.5)

98. Secondary Outcome: Cohort 3: Minimum Observed Concentration (Cmin) of Digoxin in Plasma
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Picograms per milliliter
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Picograms per milliliter | 44.127 [34.943 to 55.723] | 77.447 [60.937 to 98.430]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.755, 90% CI 2-sided [1.304 to 2.363]

99. Secondary Outcome: Cohort 3: T1/2 of Digoxin in Plasma
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours | 39.367 [37.263 to 41.589] | 32.777 [30.975 to 34.683]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 0.833, 90% CI 2-sided [0.769 to 0.902]

100. Secondary Outcome: Cohort 3: Vz/F of Digoxin in Plasma
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Liters | 923.75 [810.79 to 1052.46] | 688.49 [602.73 to 786.46]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 0.745, 90% CI 2-sided [0.653 to 0.850]

101. Secondary Outcome: Cohort 3: CL/F of Digoxin in Plasma
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Liters per Hour
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Liters per Hour | 16.26 [14.51 to 18.23] | 14.51 [12.91 to 16.31]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 0.892, 90% CI 2-sided [0.782 to 1.018]

102. Secondary Outcome: Cohort 3: Cmin of Midazolam in Plasma
Description: as for outcome 16
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Nanograms per milliliter | 0.192 [0.157 to 0.234] | 0.222 [0.181 to 0.273]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.157, 90% CI 2-sided [0.876 to 1.528]

103. Secondary Outcome: Cohort 3: T1/2 of Midazolam in Plasma
Description: as for outcome 16
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Hours
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Hours | 5.320 [4.702 to 6.018] | 6.075 [5.358 to 6.887]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 1.142, 90% CI 2-sided [1.016 to 1.283]

104. Secondary Outcome: Cohort 3: Vz/F of Midazolam in Plasma
Description: as for outcome 16
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Liters | 615.36 [537.88 to 704.01] | 371.24 [323.51 to 426.01]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 0.603, 90% CI 2-sided [0.521 to 0.699]

105. Secondary Outcome: Cohort 3: CL/F of Midazolam in Plasma
Description: as for outcome 16
Time Frame: as for outcome 16
Population: Pharmacokinetic Parameter Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Liters per Hour
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Liters per Hour | 80.17 [67.66 to 94.99] | 42.16 [35.47 to 50.10]
Statistical Analysis 1: Comparison: Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg vs Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg; Test type: Other; Ratio of Geometric LS mean = 0.526, 90% CI 2-sided [0.448 to 0.618]

106. Secondary Outcome: Cohort 3: Ae Total of Gepotidacin in Urine Following Two 3000 mg Doses (First Dose + Second Dose )
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. Ae total was calculated by adding all the fractions of drug collected over all the allotted time intervals.
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-14 Hours, 14-16 Hours, 16-18 Hours, 18-20 Hours, 20-24 Hours, 24-36 Hours, 36-48 Hours, 48-60 Hours post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Milligrams | 1066.21 (40.4)

107. Secondary Outcome: Cohort 3: Amount of Drug Excreted in Urine in a Time Interval (Ae[t1-t2]) of Gepotidacin Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 58
Time Frame: as for outcome 106
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Milligrams
  Ae (0-2), n=17: number analyzed (Participants) | 17
  Ae (0-2), n=17 | NA (NA) — NA indicates that data was not available as urine concentrations were below the lower limit of quantification. Hence, data was not calculated.
  Ae (2-4), n=18 | 117.61 (101.7)
  Ae (4-6), n=16: number analyzed (Participants) | 16
  Ae (4-6), n=16 | 103.11 (57.3)
  Ae (6-8); n=16: number analyzed (Participants) | 16
  Ae (6-8); n=16 | 70.98 (53.7)
  Ae (8-12), n=18 | 67.42 (44.3)
  Ae (12-14), n=17: number analyzed (Participants) | 17
  Ae (12-14), n=17 | 64.49 (94.1)
  Ae (14-16), n=15: number analyzed (Participants) | 15
  Ae (14-16), n=15 | 142.36 (142.3)
  Ae (16-18), n=14: number analyzed (Participants) | 14
  Ae (16-18), n=14 | 146.89 (59.4)
  Ae (18-20), n=15: number analyzed (Participants) | 15
  Ae (18-20), n=15 | 93.05 (83.5)
  Ae (20-24), n=17: number analyzed (Participants) | 17
  Ae (20-24), n=17 | 74.44 (93.9)
  Ae (24-36), n=18 | 70.01 (105.0)
  Ae (36-48); n=18 | 20.16 (46.4)
  Ae (48-60), n=18 | 8.51 (42.7)

108. Secondary Outcome: Cohort 3: AUC(0-tau) of Gepotidacin in Urine Following Two 3000 mg Doses (First Dose + Second Dose)
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis.
Time Frame: as for outcome 106
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours*micrograms per milliliter | 4770.8 (55.2)

109. Secondary Outcome: Cohort 3: AUC(0-24) of Gepotidacin in Urine Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 108
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-14 Hours, 14-16 Hours, 16-18 Hours, 18-20 Hours, 20-24 Hours post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours*micrograms per milliliter | 14333.9 (59.2)

110. Secondary Outcome: Cohort 3: AUC (0-48) of Gepotidacin in Urine Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 108
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-14 Hours, 14-16 Hours, 16-18 Hours, 18-20 Hours, 20-24 Hours, 24-36 Hours, 36-48 Hours post-dose in each Treatment Periods 1 and 2
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Hours*micrograms per milliliter | 16682.1 (59.4)

111. Secondary Outcome: Cohort 3: Percentage of the Given Dose of Drug Excreted in Urine (fe%) Following Two 3000 mg Doses of Gepotidacin (First Dose + Second Dose )
Description: as for outcome 76
Time Frame: as for outcome 106
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 18
Percent dose excreted | 17.77 (40.4)

112. Secondary Outcome: Cohort 3: CLr of Gepotidacin Following Two 3000 mg Doses (First Dose + Second Dose)
Description: as for outcome 108
Time Frame: as for outcome 106
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 17
Liters per Hour | 13.19 (34.6)

113. Secondary Outcome: Cohort 3: Number of Participants With SAE and Non-SAE
Description: as for outcome 60
Time Frame: Up to 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Participants
  Any SAE | 0 | 0
  Any non-SAE | 1 | 11

114. Secondary Outcome: Cohort 3: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 78
Time Frame: Up to 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Participants
  Basophils; To Low | 0 | 0
  Basophils; To Normal or No Change | 19 | 18
  Basophils; To High | 0 | 0
  Eosinophils; To Low | 0 | 0
  Eosinophils; To Normal or No Change | 19 | 16
  Eosinophils; To High | 0 | 2
  MCH; To Low | 0 | 0
  MCH; To Normal or No Change | 19 | 18
  MCH; To High | 0 | 0
  MCV; To Low | 0 | 0
  MCV; To Normal or No Change | 18 | 18
  MCV; To High | 1 | 0
  Erythrocytes; To Low | 2 | 1
  Erythrocytes; To Normal or No Change | 17 | 17
  Erythrocytes; To High | 0 | 0
  Hematocrit; To Low | 1 | 2
  Hematocrit; To Normal or No Change | 17 | 14
  Hematocrit; To High | 1 | 2
  Hemoglobin; To Low | 0 | 1
  Hemoglobin; To Normal or No Change | 18 | 15
  Hemoglobin; To High | 1 | 2
  Leukocytes; To Low | 0 | 0
  Leukocytes; To Normal or No Change | 19 | 17
  Leukocytes; To High | 0 | 1
  Lymphocytes; To Low | 0 | 0
  Lymphocytes; To Normal or No Change | 19 | 17
  Lymphocytes; To High | 0 | 1
  Monocytes; To Low | 0 | 1
  Monocytes; To Normal or No Change | 18 | 17
  Monocytes; To High | 1 | 0
  Neutrophils; To Low | 0 | 0
  Neutrophils; To Normal or No Change | 19 | 17
  Neutrophils; To High | 0 | 1
  Platelets; To Low | 0 | 0
  Platelets; To Normal or No Change | 19 | 18
  Platelets; To High | 0 | 0

115. Secondary Outcome: Cohort 3: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 62
Time Frame: Up to 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Participants
  ALT; To Low | 0 | 0
  ALT; To Normal or No Change | 19 | 17
  ALT; To High | 0 | 1
  Albumin; To Low | 1 | 0
  Albumin; To Normal or No Change | 18 | 17
  Albumin; To High | 0 | 1
  Alk Phos; To Low | 0 | 0
  Alk Phos; To Normal or No Change | 19 | 18
  Alk Phos; To High | 0 | 0
  AST; To Low | 0 | 0
  AST; To Normal or No Change | 18 | 18
  AST; To High | 1 | 0
  Bilirubin; To Low | 0 | 0
  Bilirubin; To Normal or No Change | 19 | 18
  Bilirubin; To High | 0 | 0
  Calcium; To Low | 1 | 1
  Calcium; To Normal or No Change | 18 | 17
  Calcium; To High | 0 | 0
  Carbon Dioxide; To Low | 0 | 0
  Carbon Dioxide; To Normal or No Change | 19 | 18
  Carbon Dioxide; To High | 0 | 0
  Chloride; To Low | 0 | 0
  Chloride; To Normal or No Change | 19 | 17
  Chloride; To High | 0 | 1
  Creatine Kinase; To Low | 0 | 0
  Creatine Kinase; To Normal or No Change | 18 | 18
  Creatine Kinase; To High | 1 | 0
  Creatinine; To Low | 0 | 0
  Creatinine; To Normal or No Change | 19 | 18
  Creatinine; To High | 0 | 0
  Direct Bilirubin; To Low | 0 | 0
  Direct Bilirubin; To Normal or No Change | 19 | 18
  Direct Bilirubin; To High | 0 | 0
  Glucose; To Low | 0 | 0
  Glucose; To Normal or No Change | 19 | 18
  Glucose; To High | 0 | 0
  Magnesium; To Low | 0 | 0
  Magnesium; To Normal or No Change | 19 | 18
  Magnesium; To High | 0 | 0
  Potassium; To Low | 0 | 0
  Potassium; To Normal or No Change | 18 | 18
  Potassium; To High | 1 | 0
  Protein; To Low | 0 | 0
  Protein; To Normal or No Change | 19 | 18
  Protein; To High | 0 | 0
  Sodium; To Low | 0 | 0
  Sodium; To Normal or No Change | 19 | 18
  Sodium; To High | 0 | 0
  BUN; To Low | 0 | 1
  BUN; To Normal or No Change | 19 | 17
  BUN; To High | 0 | 0

116. Secondary Outcome: Cohort 3: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 63
Time Frame: Up to 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Participants
  Bilirubin; To Normal or No Change | 19 | 18
  Bilirubin; To Abnormal | 0 | 0
  Glucose; To Normal or No Change | 19 | 18
  Glucose; To Abnormal | 0 | 0
  Ketones; To Normal or No Change | 16 | 17
  Ketones; To Abnormal | 3 | 1
  Leukocyte Esterase; To Normal or No Change | 13 | 13
  Leukocyte Esterase; To Abnormal | 6 | 5
  Nitrite; To Normal or No Change | 19 | 18
  Nitrite; To Abnormal | 0 | 0
  Occult Blood; To Normal or No Change | 14 | 13
  Occult Blood; To Abnormal | 5 | 5
  Protein; To Normal or No Change | 16 | 16
  Protein; To Abnormal | 3 | 2
  pH; To Low | 0 | 0
  pH; To Normal or No Change | 19 | 18
  pH; To High | 0 | 0
  Specific Gravity; To Low | 0 | 0
  Specific Gravity; To Normal or No Chan | 16 | 10
  Specific Gravity; To High | 3 | 8

117. Secondary Outcome: Cohort 3: Number of Participants With Worst Case Vital Sign Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 64
Time Frame: Up to 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Participants
  DBP; To Low | 0 | 0
  DBP; To Normal or No Change | 19 | 18
  DBP; To High | 0 | 0
  SBP; To Low | 0 | 0
  SBP; To Normal or No Change | 19 | 18
  SBP; To High | 0 | 0
  Pulse rate; To Low | 0 | 0
  Pulse rate; To Normal or No Change | 19 | 18
  Pulse rate; To High | 0 | 0

118. Secondary Outcome: Cohort 3: Number of Participants With Any Increase in Maximum Post-Baseline ECG Parameter QTc Interval
Description: as for outcome 65
Time Frame: Up to 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg
Number analyzed (Participants) | 19 | 18
Participants
  QTcB Interval | 2 | 5
  QTcF Interval | 0 | 0

119. Secondary Outcome: Cohort 4: T1/2 of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Hours | 12.848 (28.5) | 12.540 (14.2)

120. Secondary Outcome: Cohort 4: Vz/F of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Liters | 1246.70 (38.8) | 1329.83 (17.7)

121. Secondary Outcome: Cohort 4: CL/F of Gepotidacin Following Single Dose of 1500 mg in Plasma
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted
Number analyzed (Participants) | 11 | 11
Liters per Hour | 67.26 (15.5) | 73.50 (13.3)

122. Secondary Outcome: Cohort 4: Tlag of Gepotidacin in Plasma After the First Dose of 3000 mg (First Dose)-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Hours | 0 [0 to 0]

123. Secondary Outcome: Cohort 4: Vz/F of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 10
Liters | 1251.05 (34.5)

124. Secondary Outcome: Cohort 4: CL/F of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose)-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 10
Liters per Hour | 68.83 (13.9)

125. Secondary Outcome: Cohort 4: T1/2 of Gepotidacin in Plasma Following Two 3000 mg Doses (First Dose + Second Dose )-Fed State
Description: as for outcome 2
Time Frame: as for outcome 27
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 10
Hours | 12.599 (36.6)

126. Secondary Outcome: Cohort 4: Ae Total of Gepotidacin Following Single Dose of 1500 mg Under Fed Condition in Urine
Description: as for outcome 106
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed
Number analyzed (Participants) | 11
Milligrams | 293.50 (29.0)

127. Secondary Outcome: Cohort 4: Ae(t1-t2) of Gepotidacin Following Single Dose of 1500 mg Under Fed Condition in Urine
Description: as for outcome 58
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed
Number analyzed (Participants) | 11
Milligrams
  Ae (0-2) | NA (NA) — NA indicates that data was not available as urine concentrations were below the lower limit of quantification. Hence, data was not calculated
  Ae (2-4) | 102.23 (25.2)
  Ae (4-6) | 60.05 (57.0)
  Ae (6-8) | 31.61 (48.9)
  Ae (8-12) | 16.51 (97.0)
  Ae (12-24) | 17.16 (49.3)
  Ae (24-36) | 5.72 (196.5)
  Ae (36-48) | 4.28 (63.2)

128. Secondary Outcome: Cohort 4: AUC(0-24) of Gepotidacin Following Single Dose of 1500 mg Under Fed Condition in Urine
Description: as for outcome 108
Time Frame: as for outcome 55
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | 2142.4 (53.5)

129. Secondary Outcome: Cohort 4: AUC(0-48) of Gepotidacin Following Single Dose of 1500 mg Under Fed Condition in Urine
Description: as for outcome 108
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | 2293.7 (53.2)

130. Secondary Outcome: Cohort 4: Percentage of the Given Dose of Drug Excreted in Urine (fe%) for Gepotidacin 1500 mg Under Fed Condition
Description: Urine samples were collected at indicated time points. Pharmacokinetic analysis of gepotidacin was conducted using standard non-compartmental analysis. fe% was calculated as: (Ae total divided by Dose) multiplied by 100%.
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed
Number analyzed (Participants) | 11
Percent dose excreted | 19.57 (29.0)

131. Secondary Outcome: Cohort 4: CLr of Gepotidacin Following Single Dose of 1500 mg Under Fed Condition
Description: as for outcome 108
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed
Number analyzed (Participants) | 11
Liters per Hour | 13.42 (31.9)

132. Secondary Outcome: Cohort 4: Ae Total of Gepotidacin in Urine Following Two 3000 mg Doses-Fed State
Description: as for outcome 106
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-14 Hours, 14-16 Hours, 16-18 Hours, 18-20 Hours, 20-24 Hours, 24-36 Hours, 36-48 Hours, 48-60 Hours post-dose in Treatment Period 3
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Milligrams | 1334.42 (25.4)

133. Secondary Outcome: Cohort 4: Ae(t1-t2) of Gepotidacin in Urine Following Two 3000 mg Doses-Fed State
Description: as for outcome 58
Time Frame: as for outcome 132
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Milligrams
  Ae (0-2); n=11 | NA (NA) — NA indicates that data was not available as urine concentrations were below the lower limit of quantification. Hence, data was not calculated.
  Ae (2-4); n=10: number analyzed (Participants) | 10
  Ae (2-4); n=10 | 221.19 (56.7)
  Ae (4-6); n=11 | 103.68 (70.6)
  Ae (6-8); n=11 | 67.58 (49.5)
  Ae (8-12); n=11 | 65.06 (22.7)
  Ae (12-14); n=11 | 112.83 (66.3)
  Ae (14-16); n=11 | 174.62 (85.2)
  Ae (16-18); n=11 | 136.66 (68.1)
  Ae (18-20); n=11 | 90.81 (25.4)
  Ae (20-24); n=11 | 80.54 (20.4)
  Ae (24-36); n=11 | 57.62 (42.9)
  Ae (36-48); n=11 | 14.47 (36.9)
  Ae (48-60); n=10: number analyzed (Participants) | 10
  Ae (48-60); n=10 | 9.67 (61.7)

134. Secondary Outcome: Cohort 4: AUC(0-tau) of Gepotidacin in Urine Following Two 3000 mg Doses-Fed State
Description: as for outcome 108
Time Frame: as for outcome 132
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 10
Hours*micrograms per milliliter | 4996.9 (64.4)

135. Secondary Outcome: Cohort 4: AUC(0-24) of Gepotidacin in Urine Following Two 3000 mg Doses-Fed State
Description: as for outcome 108
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-14 Hours, 14-16 Hours, 16-18 Hours, 18-20 Hours, 20-24 Hours post-dose in Treatment Period 3
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 10
Hours*micrograms per milliliter | 14729.5 (59.3)

136. Secondary Outcome: Cohort 4: AUC(0-48) of Gepotidacin in Urine Following Two 3000 mg Doses-Fed State
Description: as for outcome 108
Time Frame: Pre-dose, 0-2 Hours, 2-4 Hours, 4-6 Hours, 6-8 Hours, 8-12 Hours, 12-14 Hours, 14-16 Hours, 16-18 Hours, 18-20 Hours, 20-24 Hours, 24-36 Hours, 36-48 Hours post-dose in Treatment Period 3
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 10
Hours*micrograms per milliliter | 15768.2 (58.8)

137. Secondary Outcome: Cohort 4: Percentage of the Given Dose of Drug Excreted in Urine (fe%) of Gepotidacin Following Two 3000 mg Doses-Fed State
Description: as for outcome 76
Time Frame: as for outcome 132
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Percent dose excreted | 22.24 (25.4)

138. Secondary Outcome: Cohort 4: CLr of Gepotidacin Following Two 3000 mg Dose-Fed State
Description: as for outcome 108
Time Frame: as for outcome 132
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour
Arm/Group | Cohort 4: Gepotidacin 3000 mg Fed
Number analyzed (Participants) | 11
Liters per Hour | 14.61 (19.3)

139. Other Pre Specified Outcome: Cohort 4: AUC(0-tau) of Gepotidacin Following Single Dose of 1500 mg Under Fed Condition in Urine
Description: Urine samples were collected at indicated time points. AUC(0-tau) can be calculated only for multiple doses and not for single dose as tau refers to the dosing interval. Hence, AUC(0-tau) could not be calculated for Gepotidacin 1500 mg single dose as mentioned in Reporting and Analysis Plan. The results for this outcome measure will never be posted.
Time Frame: as for outcome 54
Population: Pharmacokinetic Parameter Population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Cohort 4: Gepotidacin 1500 mg Fed
Number analyzed (Participants) | 11
Hours*micrograms per milliliter | NA (NA) — NA indicates that data was not available as AUC(0-tau) could not be calculated for single dose as it can be calculated only for multiple doses.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and non-serious adverse events (non-SAE) were collected up to 17 days during Cohort 1; up to 26 days during Cohort 2; up to 30 days during Cohort 3 and up to 22 days during Cohort 4.
Description: Safety Population comprised of all participants who took at least 1 dose of study intervention. Participants with adverse events that occurred during Days 1 to 7 in Period 2 after the exposure of Rifampicin 600 mg and those occurred during Days 8 to 9 in Period 2 after exposure of Gepotidacin 1500 mg + Rifampicin 600 mg were summarized separately. Only those participants with data available at specified time points were analyzed.
Arm/Group | Cohort 1: Gepotidacin 1500 mg | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg | Cohort 2: Period 1: Gepotidacin 1500 mg | Cohort 2: Period 2 (Days 1 to 7) Rifampicin 600 mg | Cohort 2: Period 2 (Days 8 to 9) Gepotidacin 1500 mg + Rifampicin 600 mg | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg | Cohort 4: Placebo | Cohort 4: Gepotidacin 1500 mg Fed | Cohort 4: Gepotidacin 1500 mg Fasted | Cohort 4: Gepotidacin 3000 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/17 | 0/17 | 0/14 | 0/19 | 0/18 | 0/3 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/17 | 0/17 | 0/14 | 0/19 | 0/18 | 0/3 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 3/17 | 2/17 | 2/14 | 1/19 | 11/18 | 0/3 | 1/11 | 2/11 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Gepotidacin 1500 mg (N=14) | Cohort 1: Gepotidacin 1500 mg + Cimetidine 400 mg (N=13) | Cohort 2: Period 1: Gepotidacin 1500 mg (N=17) | Cohort 2: Period 2 (Days 1 to 7) Rifampicin 600 mg (N=17) | Cohort 2: Period 2 (Days 8 to 9) Gepotidacin 1500 mg + Rifampicin 600 mg (N=14) | Cohort 3: Digoxin 0.5 mg + Midazolam 2 mg (N=19) | Cohort 3:Gepotidacin 3000 mg + Digoxin 0.5 mg + Midazolam 2 mg (N=18) | Cohort 4: Placebo (N=3) | Cohort 4: Gepotidacin 1500 mg Fed (N=11) | Cohort 4: Gepotidacin 1500 mg Fasted (N=11) | Cohort 4: Gepotidacin 3000 mg Fed (N=11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT04493931/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT04493931/SAP_001.pdf